CLINICAL TRIAL: NCT04752579
Title: Effects of a Mat Pilates Exercise Program on Pain, Functional Ability and Balance in Elderly Women With Chronic Nonspecific Low Back Pain
Brief Title: Effects of a Mat Pilates Exercise Program on Elderly Women With Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, LYTRAS DIMITRIOS, Dimitrios Lytras PT, PhD, Postdoctoral Research Fellow Affiliation: Aristotle University of Thessaloniki, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-48/2021
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Low Back Pain
Keywords: Mat-pilates exercises; elderly; chronic low back pain; physical therapy; rehabilitation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: A masked assessor conducted the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise program (Experimental): Participants allocated to this group will receive a 10-week Pilates exercise program with each session having a duration of 45'.
  Interventions: Other: Pilates exercise program
- Control (Placebo Comparator): Participants allocated to this group received general consulting instructions and a home-based general exercise sheet
  Interventions: Other: Pilates exercise program

INTERVENTIONS:
Other: Pilates exercise program — The program will be individually supervised and will be conducted twice a week at the physiotherapy center.
  • Slow execution of 7-10 repetitions of the following Pilates exercises: Pelvic Curl, Pilates Single Legs Lifts & Leg Change, Twist Supine Pilates exercise, Chest Lifts Pilates Exercise, Chest Lift with Rotation Pilates exercise, 100's Prep Pilates Exercise, Single Leg Stretch Pilates Exercise, Front Support Pilates Exercise and Basic Back Extension Pilates Exercise. After the 6th week, while the person will be familiar with the basic exercises of the Pilates method the following exercises will be added: Leg Pull Front, Side Bend Pilates Exercise, Sphinx - Abdominal Lift Pilates Exercise, Shoulder Bridge Prep Pilates and Shoulder Bridge Pilates Exercise. Each session will be completed with breathing exercises and stretching exercises of the torso and lower limbs for 5 minutes.

SUMMARY:
The technique of Pilates exercises on a mat has proven to be effective and practically applicable to patients with chronic back pain. However, its application in women over 65 years has not been adequately studied.

Objective: This assessor-blind randomized clinical trial aims to study the effect of a mat Pilates exercise program on pain and functional ability of elderly women with chronic nonspecific low back pain.

Methods: 60 elderly women with chronic nonspecific low back pain (duration of symptoms more than 12 weeks) are expected to participate in this study. Participants will be divided into two groups of 30 people each; one being intervention and one control. The intervention group will follow a custom mat Pilates program (twice per week) for 10 weeks, while the control group will not follow any treatment. Pain, functionality, balance, the number of painkillers administered, and adherence to exercise will be assessed at the beginning and end of the study and will be re-examined six months later.

DETAILED DESCRIPTION:
The technique of Pilates exercises on a mat has proven to be effective and practically applicable to patients with chronic back pain. However, its application in women over 65 years has not been adequately studied.

Objective: This assessor-blind randomized clinical trial aims to study the effect of a mat Pilates exercise program on pain and functional ability of elderly women with chronic nonspecific low back pain.

Methods: 60 non-active elderly women with chronic nonspecific low back pain (duration of symptoms more than 12 weeks) are expected to participate in this study. Participants will be divided into two groups of 30 people each; one being intervention and one control. The intervention group will follow a custom mat Pilates program (twice per week), while the control group will not follow any treatment. Primary outcomes will include pain with the visual analog scale for pain and functionality with the Roland-Morris Questionnaire (RMQ). Secondary outcomes will include the balance with the Berg balance scale and the Timed Up and Go test, the number of painkillers administered, and the adherence to the exercise that will be evaluated at the beginning and at the end of the study and re-evaluated six months after the end of the intervention. The treatment period will be 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of chronic back pain lasting more than 12 weeks
* Score on the Visual Analog Scale for pain less than 70mm
* Timed Up and Go test score less than 15sec

Exclusion Criteria:

* Low back pain due to a serious pathology that refers to a red flag such as malignancy, vertebral fracture, osteomyelitis, rheumatoid arthritis, Cauda Equina Syndrome (CES)
* Participation in another exercise program in the last six months
* Diagnosed with neurodegenerative disease (e.g., Parkinson's disease)
* Recent stroke
* Senile dementia

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Female
Enrollment: 63 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in Low back pain intensity with the Visual Analogue Scale (VAS) | pre-treatment, Week: 10, 6-month follow-up
  VAS is a card with an uncalibrated scale ranging from 0-100mm on the one side with each millimeter representing one pain level (0 representing no pain and 100 representing the worst pain in life). The patient subjectively estimated their pain level by marking a vertical line on the uncalibrated scale between 0 and 100.
  Then the exact value of pain intensity could be obtained with a single ruler. Hence, the higher the value, the more intense the pain. VAS is widely used as it is easy to implement and is characterized by good psychometric propert
Changes in Roland Morris Disability Questionnaire | pre-treatment, Week: 10, 6-month follow-up
  Disability associated with low back pain in the last 24 hours will be assessed using the Greek version of the Roland Morris Disability Questionnaire (Boscainos et al., 2003). This questionnaire has showed good test -retest reliability with intraclass correlation (ICC) ranging from 0.42 to 0.91 (Macedo et al., 2010), while Boscainos (2003), reports that the internal consistency reliability for the Greek version reached a Cronbach's alpha coefﬁcient of 0.885. This questionnaire consists of 24 items that are related to daily activities which patients often report difficulty performing due to low back pain. Every positive answer earns a point and the final score is calculated by adding all the points. Thus, the higher the score is, the greater the limitation (Stratford, 1996).
Changes in Timed Up and Go (TUG) Test | pre-treatment, Week: 10, 6-month follow-up
  The TUG test is a performance-based measure of functional mobility that was initially developed to identify mobility and dynamic balance impairments in older adults (Cameron and Monroe, 2007; Swearingen and Brach, 2001; Podsiadlo and Richardson, 1991). The TUG test has demonstrated high interrater and intrarater reliability when used to examine elderly adults (Cameron and Monroe, 2007; Swearingen and Brach, 2001). The test requires the subject to rise from a chair, walk three meters at a comfortable pace to a mark placed on the floor, turn around, walk back to the starting point, and return to sitting on the chair. The test's score is the time it takes the subject to complete the test.
Changes in Berg Balance Scale | pre-treatment, Week: 10, 6-month follow-up
  The Berg balance scale is a tool suggested by Berg (Berg et al., 1989; Berg et al., 1992) to evaluate balance in the elderly. The test involves performing 14 tests of gradually increasing difficulty where in each one, the subject is asked to maintain a given position for a specific time or conduct specific tasks. Each of the 14 tests on the list is graded according to the balancing ability of the examinee from 0 to 4 points (with 0 indicating low balance ability while 4 high). Accord to Berg et al. (1992), a score of 56 indicates functional balance whereas a score lower than 45 indicates notable balance deficits, which have been related to increased fall risk.

SECONDARY OUTCOMES:
Changes in the number of pills consumed via Pill Consumption Log | pre-treatment, Month: 1,3,6, post-intervention
  Participants will be asked to write down in a special diary the number of pills administered (anti-inflammatory and/or painkillers) during the follow-up period. The log will be kept kept on a weekly basis and the assessor will collect the data by phone 2-3 times a month.
Changes in adherence to exercise via Exercise Diary keeping | Time Frame: pre-treatment, Month: 1,3,6, post-intervention
  After the ten weeks the participants of both groups will be asked to perform the specific exercise programs twice per week for a period of three months recording the adherence or not to the exercise programs in a weekly diary while the assessor will collect the data by phone 2-3 times a month.

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Sykaras, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Department of Physical Education and Sports Sciences, Thessaloniki, Thermi, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lytras D, Iakovidis P, Sykaras E, Kottaras A, Kasimis K, Myrogiannis I, Barouxakis A, Tarfali G. Effects of a tailored mat-Pilates exercise program for older adults on pain, functioning, and balance in women with chronic non-specific low back pain: a randomized controlled trial. Aging Clin Exp Res. 2023 Dec;35(12):3059-3071. doi: 10.1007/s40520-023-02604-7. Epub 2023 Nov 7. PMID 37934400